CLINICAL TRIAL: NCT03856242
Title: Benign Prostatic Hyperplasia and Ischemic Heart DIsease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Vinarov Andrey, Professor, I.M. Sechenov First Moscow State Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-19
Record Dates: First submitted 2019-02-24; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Ischaemic Heart Disease (IHD); Benign Prostatic Hyperplasia (BPH); Lower Urinary Tract Symptoms (LUTS)
MeSH Terms: conditions — Coronary Artery Disease; Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Tamsulosin; Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No intervention (No Intervention): It included the patients in whom during urination certain changes in HM were registered. The Group 1 patients' age varied from 63 to 79 years (mean 68.6±4.94 years). Nearly all except two patients (cardiac background of these patients did not require medical or surgical correction) from this group received cardiotropic therapy which did not change during one-month follow-up.
- Tamsulosin (Active Comparator): This group enrolled 28 patients in whom primary HM detected certain alterations (VE, SVE, ST segment depression) which did not coincide with the act of urination. The age of patients was from 57 to 81 years (mean 71.3±1.1 years). In order to improve impaired urination were also received Tamsulosin at a dose of 0.4 mg once daily (in the morning) for the whole period of follow up and treatment. Tamsulosin Oral Capsule.
  Interventions: Drug: Tamsulosin Oral Capsule
- TURP (Active Comparator): This group was composed of patients for whom after examination for symptoms of IHD and LUTS/BPH a decision was made on the necessity to perform operative treatment of BPH. TURP operation was indicated due to pronounced urination disorders which were most important amongst the patient's complaints. The patients' age varied from 59 to 77 years (mean 67.5±2.1 years).
  Interventions: Procedure: TURP

INTERVENTIONS:
Drug: Tamsulosin Oral Capsule — Tamsulosin Oral Capsule - alpha-1-adrenoblocker for treatment LUTS/BPH 0.4 mg
  Other Names: Tamsulosin
  Arms: Tamsulosin
Procedure: TURP — Routine transurethral prostatic resection
  Arms: TURP

SUMMARY:
To examine the dynamics of 24 - hours ECG monitoring parameters (Holter monitoring) in patients with ischaemic heart disease (IHD) before and after treatment of voiding dysfunctions resulted from benign prostatic hyperplasia (BPH) with the indications for either conservative or operative treatment.

A total of eighty-three 57-to-81-year-old (mean age 70.4±5.75 years) patients with BPH and accompanying IHD were examined at the Institute of Urology and Human Reproductive Health and Clinic of Cardiology of the Sechenov University.

DETAILED DESCRIPTION:
A total of eighty-three 57-to-81-year-old (mean age 70.4±5.75 years) patients diagnosed with BPH and accompanying IHD were examined at the Institute of Urology and Human Reproductive Health and Clinic of Cardiology of the Sechenov University.

Depending on the results of primary Holter monitoring (HM) and the method of correction (medicamentous or operative) of LUTS/BPH, all patients were subdivided into 3 groups:

Group 1 (n=20) included patients in whom primary HM revealed ECG alterations appearing or deteriorating during urination; all these patients along with recommended cardiotropic therapy, for improving impaired urination received tamsulosin at a dose of 0.4 mg once daily (in the morning) for the whole period of follow-up and treatment.

Group 2 (n=28) was composed of patients who had Holter-detected diagnostically significant ECG alterations, however, nonrelated to the act of urination; all these patients, along with the recommended cardiac therapy, in order to improve impaired urination were also received tamsulosin at a dose of 0.4 mg once daily (in the morning) for the whole period of follow up and treatment.

Group 3 (n=35) consisted of patients with BPH and IHD found to have pronounced impairments severe obstructed urination and transurethral resection of the prostate (TURP) was performed. Like in the previous group HM demonstrated diagnostically significant changes in the ECG, not however related to the act of urination.

Criteria for inclusion into the study: 1) patient's consent; 2) absence of severe accompanying pathology hampering carrying out the study (mental disorders, musculoskeletal system diseases, oncological diseases); 3) LUTS/BPH, with the total score by the IPSS more than or equal to 8; 4) functional class II-IV angina of effort; 5) non-ST segment depression postinfarction cardiosclerosis.

Exclusion criteria: 1) presence of cystostomic drainage; 2) long-term medicamentous therapy of prostatic hyperplasia (alpha-adrenoblockers, 5-alpha-reductase inhibitors and others) - for the groups of patients of conservative treatment of BPH; 3) patients after operative treatment of prostatic hyperplasia (TUR of prostatic hyperplasia, transvesical adenomectomy, etc.); 4) urinary bladder stones; 5) acute urinary retention; 6) "paradoxical" ischuria; 7) changes on the ECG hampering its interpretation (complete left bundle branch block, cicatricial changes after endured myocardial infarction, permanent form of ciliary arrhythmia); 8) acute forms of ischaemic heart disease.

Criteria for withdrawal: voluntary refusal of the patient from further follow up;

Beside interviewing (in the presence of angina, the patients filled in the Seattle Angina Questionnaire), the patients were subjected to measuring arterial pressure on both arms, biochemical blood analysis (measuring the level of triglycerides, cholesterol, if necessary, high-, low- and very-low density lipoproteins), standard 12-lead ECG. All patients in order to verify the diagnosis of IHD underwent detailed examination in the settings of a cardiological hospital including, if required, the following studies: tread-mill, stress-echocardiography, coronarography, multispiral computed tomography of the coronary arteries.

The severity of BPH symptoms and quality of life of patients were assessed by means of the IPSS and QoL questionnaires. Uroflowmetry was used to determine the degree of impairments of urination. Besides, to specify the dimensions of the prostate, its volume and to measure the amount of residual urine investigators performed transabdominal ultrasound examination (if necessary also transcatheter ultrasound), as well as digital rectal examination and blood analysis for PSA and, if indicated, biopsy of the prostate to rule out cancerous prostatic lesion.

The key method in the study was 24-hour ECG (Holter) monitoring using the Schiller MT 200 device (Switzerland). Deciphering the data of 24-hour ECG monitoring, investigators examined the dynamics of the ST segment and changes in the cardiac rhythm during urination, which was registered by the patient by depressing the respective button on the device and keeping a diary, and totally during the whole period (24 hours) of Holter monitoring.

Then, some patients (n=48) received therapy with tamsulosin for 30 days at a dose of 0.4 mg at night, and others (n=35) underwent TUR for prostatic hyperplasia. After a month on the background of continuing cardiac therapy and administration of tamsulosin in the group of conservative treatment investigators evaluated the subjective symptomatology by the IPSS and QoL scales, performed uroflowmetry, ultrasound examination of the prostate and the volume of residual urine, standard ECG and repeat 24-hour ECG monitoring with registering the time of urination. If necessary, the patients filled in the Seattle Angina Questionnaire again.

All procedures performed in the study were in accordance with standard clinical care and were in accordance with the ethical standards of the institutional and/or national research committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards.

Study was approved by Sechenov University IRB. Informed consent was obtained from all individual participants included in the study.

The data were processed using the methods of descriptive statistics, Student's t-test for paired values, in the programme BIOSTAT.

ELIGIBILITY:
Inclusion Criteria:

* LUTS/BPH, with the total score by the IPSS more than or equal to 8;
* Functional class II-IV angina of effort;
* Non-ST segment depression postinfarction cardiosclerosis.

Exclusion Criteria:

* Presence of cystostomic drainage;
* Long-term LUTS/BPH therapy of prostatic hyperplasia (alpha-adrenoblockers, 5-alpha-reductase inhibitors and others) - for the groups of patients of conservative treatment of BPH;
* Patients after operative treatment of prostatic hyperplasia (TUR of prostatic hyperplasia, transvesical adenomectomy, etc.);
* Urinary bladder stones;
* Acute urinary retention;
* Changes on the ECG hampering its interpretation (complete left bundle branch block, cicatricial changes after endured myocardial infarction, permanent form of ciliary arrhythmia);
* Acute forms of ischaemic heart disease.

Ages: 57 Years to 81 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Benign prostatic hyperplasia - is a disease diagnosed only in males older than 50 years
Enrollment: 83 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Changes from the baseline 24 - hours ECG monitoring parameters (Holter monitoring) in patients with ischaemic heart disease (IHD) before and after treatment of voiding dysfunctions. | up to 6 months
  Changes of the ST segment and of the cardiac rhythm during urination, which was registered by the patient by depressing the respective button on the device and keeping a diary, and totally during the whole period (24 hours) of Holter monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Z Vinarov, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University

REFERENCES:
- [Derived] Fiev DN, Vinarov AZ, Tsarichenko DG, Kopylov PY, Demidko YL, Syrkin AL, Rapoport LM, Alyaev YG, Glybochko PV. Holter Monitoring (24-Hour ECG) Parameter Dynamics in Patients with Ischemic Heart Disease and Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia. Adv Ther. 2019 Aug;36(8):2072-2085. doi: 10.1007/s12325-019-00977-8. Epub 2019 May 30. PMID 31148056